CLINICAL TRIAL: NCT00369330
Title: Prospective, Randomized Parallel-group Study for Evaluation of Impact of Early Versus Delayed Cardioversion of Acute Atrial Fibrillation on Further Clinical Course
Brief Title: KONVERT-AF - Relevance of Point in Time for Conversion of Acute Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn because of insufficient financial capacities
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFNET-B03
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2006-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; early cardioversion; electrical cardioversion
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Device: external electrical cardioversion

SUMMARY:
To investigate if in acute symptomatic atrial fibrillation (AF) the early (>2 hrs but within 12 hrs of the beginning of the arrhythmia) electrical cardioversion leads to a longer recurrence-free interval than the delayed cardioversion (> 36 hrs but < 48 hrs after the beginning of the arrhythmia) within the first 3 months after cardioversion.

DETAILED DESCRIPTION:
So far it is unknown if early or delayed cardioversion is most beneficial for patient outcome and which strategy is best to prevent recurrence of AF. The KONVERT-AF trial investigates if in acute symptomatic AF the early (>2 hrs but within 12 hrs of the beginning of the arrhythmia) electrical cardioversion leads to a longer recurrence-free interval than the delayed cardioversion (> 36 hrs but < 48 hrs after the beginning of the arrhythmia) within the first 3 months after cardioversion. Primary endpoint is the time to the first recurrence of AF. The KONVERT-AF trial will be conducted as prospective, randomized, non-blinded multicentre study. It is planned to include 380 patients in 10-20 recruitment centres.

ELIGIBILITY:
Inclusion Criteria:

* documented AF that began between 2 and 8 hrs before randomization
* indication for electrical cardioversion.
* age above 18 yrs
* written informed consent

Exclusion Criteria:

* AF caused by not adequately treated reversible conditions(e.g. myocardial infarction, thyrotoxicosis, ethanol intoxication, infection, pericarditis, surgery)
* newly initiated (i.e. within 7 days before randomization) antiarrhythmic agents of class I, II and/or III
* catheter ablation of AF within 3 months before randomization
* pacemaker or icd
* myocardial infarction within 3 months before randomization
* urgent need to cardioversion of AF because of associated potentially dangerous symptoms such as chest pain, syncope, dyspnea
* contraindications for therapy with vitamin k-antagonists
* intracardial thrombus
* primary indication for pharmacological cardioversion
* in females: pregnancy, lactation period or no sufficient contraception within last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09

SECONDARY OUTCOMES:
Number of electrical cardioversion because of AF
Need to initiate or change medical antiarrhythmic treatment because of recurrence of AF
Number and length of stay of hospitalization because of cardiovascular reasons
Number of thromboembolic events
Number of therapy non-responder and early recurrence of AF
AF burden

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Lewalter, MD, Principal Investigator — Medizinische Klinik und Poliklinik II - Universitätsklinikum Bonn, Bonn, Germany
Locations (1):
- Medizinische Klinik und Poliklinik II, University Hospital of Bonn, Bonn, Germany

REFERENCES:
- See also: Homepage of german atrial fibrillation network — http://www.kompetenznetz-vorhofflimmern.de